CLINICAL TRIAL: NCT00094614
Title: A Randomized Trial Comparing Daily Atropine Versus Weekend Atropine
Brief Title: Trial Comparing Daily Atropine Versus Weekend Atropine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEI-94; 2U10EY011751 (NIH)
Record Dates: First submitted 2004-10-21; First posted 2004-10-22 (Estimated); Last update posted 2010-03-25 (Estimated); Status verified 2006-04

CONDITIONS: Amblyopia
MeSH Terms: conditions — Amblyopia | interventions — Atropine

INTERVENTIONS:
Drug: Atropine

SUMMARY:
The goals of this study are:

* To compare the visual acuity outcome in the amblyopic eye after 17 weeks of daily use of atropine versus weekend-only use of atropine.
* To compare the proportion of patients achieving a complete treatment response (defined as amblyopic eye acuity >20/25 or equal to that of the sound eye in the absence of a reduction in the sound eye acuity from baseline) with daily atropine versus weekend-only atropine.

DETAILED DESCRIPTION:
Amblyopia is the most common cause of monocular visual impairment in both children and young and middle-aged adults. Patching has been the mainstay of amblyopia therapy. It is generally held that the response to treatment is best when it is instituted at an early age and is poor when attempted after eight years of age.

The study 'Occlusion versus Pharmacologic Therapy for Moderate Amblyopia', a randomized trial of 419 children meeting entry criteria similar to the current study, found that both atropine 1% (one drop daily) and patching (6 hours to full time daily) produced visual acuity improvement of similar magnitude and that both are appropriate treatment modalities for the management of moderate amblyopia in children. Patching has the potential advantage of a more rapid improvement in visual acuity and possibly a slightly better acuity outcome, whereas atropine has the potential advantage of easier administration and lower cost.

Through its cycloplegic effect, atropine prevents accommodation, blurring the sound eye at near fixation. The blurring effect can be augmented by reducing the spectacle correction of hyperopia in the sound eye. The cycloplegic effect lasts at least partially for a week or longer. Therefore, some pediatric eye care providers believe that daily use of atropine is unnecessary and treatment may be effective at a dosage of as little as once a week. One advantage of less frequent dosing is a potential reduction in side effects, including any potential adverse effect on the vision in the sound eye (reverse amblyopia), on ocular alignment, and on binocularity. The current study will assess whether prescribing atropine once a day produces a better visual outcome than does atropine used only on the two weekend days.

In the 'Occlusion versus Pharmacologic Therapy for Moderate Amblyopia' study, the 6-month outcome data showed that more patients treated with atropine had a reduction in visual acuity of 1 or more lines in the sound eye than did patients treated with patching. Visual acuity was decreased from baseline by 1 line in 15% of the atropine group compared with 7% of the patching group and by 2 or more lines in 9% of the atropine group and 1% of the patching group. Only one patient (in the atropine group) was actively treated for a presumed treatment-related decrease in sound eye acuity, with return of acuity to its baseline level. Some of the cases of reduced acuity were unequivocally due to the use of improper refractive correction for the sound eye testing (including nine cases in which the testing was done with a plano lens prescribed for therapeutic effect rather than the proper corrective lens). In other cases, we speculated that there was a residual cycloplegic effect of atropine combined with improper refractive correction related to previously latent hyperopia becoming manifest hyperopia during the period of atropine treatment, although there were not data to fully document this in all cases. All 47 atropine group patients with a decrease of one or more lines at six months have had subsequent follow-up exams. Acuity on the subsequent testing was the same or better than that at baseline in 42 of the 47 patients: 22 while still on atropine treatment (11 with the same refractive correction and 11 with a different refractive correction) and 20 after atropine was discontinued (6 with the same refractive correction and 14 with a different refractive correction). In the other five patients, acuity on subsequent testing was decreased from baseline by one line (3 on atropine, 2 off atropine). Thus, there did not appear to be a long-term safety concern for atropine, but the data were inconclusive as to whether atropine caused an actual, though transient, treatment-related decrease in sound eye acuity. One of the objectives of the current study will be to provide additional data on the effect of atropine on the sound eye.

The study is a randomized trial comparing atropine regimes for children with moderate amblyopia. It will consist of about 160 children. Patients in the daily atropine group receive atropine 1% one drop daily in the sound eye. Patients in the weekend atropine group will receive atropine 1% twice a week (Saturday and Sunday) in the sound eye. Visual acuity is the major study outcome. It is measured after 17 weeks of treatment with either daily or weekend atropine.

ELIGIBILITY:
Inclusion Criteria:

* Age < 7 years
* Able to measure surrounded single optotype visual acuity using the ATS single-surround HOTV protocol (this will in effect exclude all patients <2 years old and many <3 years old)
* Amblyopia associated with strabismus, anisometropia, or both
* If anisometropia is present (as per protocol definition), refractive error corrected with spectacles for a minimum of 4 weeks
* Visual acuity in the amblyopic eye < 20/40 and >20/80
* Visual acuity in the sound eye > 20/40 and inter-eye acuity difference >3 logMAR lines

Exclusion Criteria:

* Amblyopia treatment (other than spectacles) in the past month and no more than one month of amblyopia treatment in the past 6 months
* Myopia more than a spherical equivalent of -6.00 D in the amblyopic eye
* Myopia more than a spherical equivalent of -0.50 D in the sound eye

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 168
Dates: Start 2002-06; Study Completion 2003-04

PRIMARY OUTCOMES:
Visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Michael X Repka, MD, Study Chair — Wilmer Eye Institute; Jonathan M Holmes, MD, Study Chair — Mayo Clinic Department of Ophthalmology
Locations (1):
- Wilmer Eye Institute, Baltimore, Maryland, United States

REFERENCES:
- [Result] Repka MX, Cotter SA, Beck RW, Kraker RT, Birch EE, Everett DF, Hertle RW, Holmes JM, Quinn GE, Sala NA, Scheiman MM, Stager DR Sr, Wallace DK; Pediatric Eye Disease Investigator Group. A randomized trial of atropine regimens for treatment of moderate amblyopia in children. Ophthalmology. 2004 Nov;111(11):2076-85. doi: 10.1016/j.ophtha.2004.04.032. PMID 15522375
- [Derived] Wallace DK, Lazar EL, Melia M, Birch EE, Holmes JM, Hopkins KB, Kraker RT, Kulp MT, Pang Y, Repka MX, Tamkins SM, Weise KK; Pediatric Eye Disease Investigator Group. Stereoacuity in children with anisometropic amblyopia. J AAPOS. 2011 Oct;15(5):455-61. doi: 10.1016/j.jaapos.2011.06.007. PMID 22108357
- [Derived] Christoff A, Repka MX, Kaminski BM, Holmes JM; Pediatric Eye Disease Investigator Group. Distance versus near visual acuity in amblyopia. J AAPOS. 2011 Aug;15(4):342-4. doi: 10.1016/j.jaapos.2011.05.004. PMID 21907115
- [Derived] Repka M, Simons K, Kraker R; Pediatric Eye Disease Investigator Group. Laterality of amblyopia. Am J Ophthalmol. 2010 Aug;150(2):270-4. doi: 10.1016/j.ajo.2010.01.040. Epub 2010 May 8. PMID 20451898